CLINICAL TRIAL: NCT00829738
Title: Pantoprazole 20/40 mg in Reflux-Associated Complaints With Focus on Gastrointestinal Symptoms
Brief Title: Efficacy of Pantoprazole 20/40 mg Once Daily (od) in Patients Older Than 12 Years Who Have Gastrointestinal Symptoms of Reflux Disease
Acronym: PARADE
Status: Completed | Type: Observational
Sponsor: Nycomed (Industry)
Responsible Party: Medical Responsible, Nycomed Deutschland GmbH
Other Study IDs: P2-9999-011-DE
Record Dates: First submitted 2009-01-13; First posted 2009-01-27 (Estimated); Results first posted 2010-09-24 (Estimated); Last update posted 2012-05-08 (Estimated); Status verified 2012-05

CONDITIONS: Gastroesophageal Reflux Disease
Keywords: PPI therapy; pantoprazole; GERD (Erosive Gastroesophageal Reflux Disease)
MeSH Terms: conditions — Gastroesophageal Reflux | interventions — Pantoprazole

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Group 1: All patients enrolled
  Interventions: Drug: Pantoprazole

INTERVENTIONS:
Drug: Pantoprazole — This was an observational study. Therefore, the physician decided about dosage according to individual needs (20 or 40 mg pantoprazole).

SUMMARY:
The aim of this study was to evaluate the effect of 14 days treatment with Pantoprazole 40 mg and 20 mg on gastroesophageal reflux disease (GERD) related symptoms in a large patient population.

ELIGIBILITY:
Main inclusion criteria:

* Outpatients with gastroesophageal reflux disease (GERD)

Main exclusion criteria:

* Criteria as defined in the Summary of Product Characteristics

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Outpatients
Sampling Method: Non-Probability Sample
Enrollment: 4188 (Actual)
Dates: Start 2009-01; Primary Completion 2009-04 (Actual); Study Completion 2009-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas D. Bethke, MD, MBA, Study Director — Nycomed Deutschland GmbH, 78467 Konstanz, Germany
Locations (551):
- Germany (551):
  - Nycomed Deutschland GmbH, Aachen
  - Nycomed Deutschland GmbH, Ahrensburg
  - Nycomed Deutschland GmbH, Alpenrod
  - Nycomed Deutschland GmbH, Altenburg
  - Nycomed Deutschland GmbH, Altenholz
  - Nycomed Deutschland GmbH, Altenkirchen
  - Nycomed Deutschland GmbH, Altflußheim
  - Nycomed Deutschland GmbH, Alzenau in Unterfranken
  - Nycomed Deutschland GmbH, Angermünde
  - Nycomed Deutschland GmbH, Anklam
  - Nycomed Deutschland GmbH, Annweiler am Trifels
  - Nycomed Deutschland GmbH, Ansbach
  - Nycomed Deutschland GmbH, Apolda
  - Nycomed Deutschland GmbH, Arnstadt
  - Nycomed Deutschland GmbH, Ascheberg
  - Nycomed Deutschland GmbH, Aschendorf
  - Nycomed Deutschland GmbH, Aschersleben
  - Nycomed Deutschland GmbH, Aue
  - Nycomed Deutschland GmbH, Augsburg
  - Nycomed Deutschland GmbH, Augustusburg
  - Nycomed Deutschland GmbH, Aumühle
  - Nycomed Deutschland GmbH, Babenhausen
  - Nycomed Deutschland GmbH, Bad Arolsen
  - Nycomed Deutschland GmbH, Bad Berka
  - Nycomed Deutschland GmbH, Bad Berleburg
  - Nycomed Deutschland GmbH, Bad Bevensen
  - Nycomed Deutschland GmbH, Bad Bramstedt
  - Nycomed Deutschland GmbH, Bad Doberan
  - Nycomed Deutschland GmbH, Bad Dürkheim
  - Nycomed Deutschland GmbH, Bad Langensalza
  - Nycomed Deutschland GmbH, Bad Liebenwerda
  - Nycomed Deutschland GmbH, Bad Oeynhausen
  - Nycomed Deutschland GmbH, Bad Oldesloe
  - Nycomed Deutschland GmbH, Bad Orb
  - Nycomed Deutschland GmbH, Bad Pyrmont
  - Nycomed Deutschland GmbH, Bad Rappenau
  - Nycomed Deutschland GmbH, Bad Salzuflen
  - Nycomed Deutschland GmbH, Bad Sassendorf
  - Nycomed Deutschland GmbH, Bad Schwalbach
  - Nycomed Deutschland GmbH, Bad Tölz
  - Nycomed Deutschland GmbH, Bad Windsheim
  - Nycomed Deutschland GmbH, Bad Winsheim
  - Nycomed Deutschland GmbH, Badel
  - Nycomed Deutschland GmbH, Bahrdorf
  - Nycomed Deutschland GmbH, Bakum
  - Nycomed Deutschland GmbH, Balingen
  - Nycomed Deutschland GmbH, Bamberg
  - Nycomed Deutschland GmbH, Barmstedt
  - Nycomed Deutschland GmbH, Bausendorf
  - Nycomed Deutschland GmbH, Bechhofen
  - Nycomed Deutschland GmbH, Beckum
  - Nycomed Deutschland GmbH, Beckum-Neubeckum
  - Nycomed Deutschland GmbH, Bergisch Gladbach
  - Nycomed Deutschland GmbH, Bergkamen
  - Nycomed Deutschland GmbH, Berlin
  - Nycomed Deutschland GmbH, Bernburg
  - Nycomed Deutschland GmbH, Berne
  - Nycomed Deutschland GmbH, Bernkastel-Kues
  - Nycomed Deutschland GmbH, Beucha
  - Nycomed Deutschland GmbH, Beverungen
  - Nycomed Deutschland GmbH, Bielefeld
  - Nycomed Deutschland GmbH, Bietigheim-Bissingen
  - Nycomed Deutschland GmbH, Birkendorf
  - Nycomed Deutschland GmbH, Birkenwerder
  - Nycomed Deutschland GmbH, Blankenhain
  - Nycomed Deutschland GmbH, Blieskastel
  - Nycomed Deutschland GmbH, Bochum
  - Nycomed Deutschland GmbH, Bonn
  - Nycomed Deutschland GmbH, Bonndorf
  - Nycomed Deutschland GmbH, Borna
  - Nycomed Deutschland GmbH, Böblingen
  - Nycomed Deutschland GmbH, Böhlen
  - Nycomed Deutschland GmbH, Brake
  - Nycomed Deutschland GmbH, Brakel
  - Nycomed Deutschland GmbH, Braunschweig
  - Nycomed Deutschland GmbH, Brausbedra
  - Nycomed Deutschland GmbH, Breidenbach
  - Nycomed Deutschland GmbH, Bremen
  - Nycomed Deutschland GmbH, Bremen-Lehe
  - Nycomed Deutschland GmbH, Bremerhaven
  - Nycomed Deutschland GmbH, Brilon
  - Nycomed Deutschland GmbH, Bröckel
  - Nycomed Deutschland GmbH, Bruchsal
  - Nycomed Deutschland GmbH, Brühl
  - Nycomed Deutschland GmbH, Brühl-Pingsdorf
  - Nycomed Deutschland GmbH, Buckow
  - Nycomed Deutschland GmbH, Burgdorf, Hanover
  - Nycomed Deutschland GmbH, Burgstädt
  - Nycomed Deutschland GmbH, Butzbach
  - Nycomed Deutschland GmbH, Büdingen
  - Nycomed Deutschland GmbH, Castrop-Rauxel
  - Nycomed Deutschland GmbH, Chemnitz
  - Nycomed Deutschland GmbH, Cismar
  - Nycomed Deutschland GmbH, Clausthal-Zellerfeld
  - Nycomed Deutschland GmbH, Claußnitz
  - Nycomed Deutschland GmbH, Coesfeld
  - Nycomed Deutschland GmbH, Cologne
  - Nycomed Deutschland GmbH, Dabel
  - Nycomed Deutschland GmbH, Darmstadt
  - Nycomed Deutschland GmbH, Deggingen
  - Nycomed Deutschland GmbH, Delitzsch
  - Nycomed Deutschland GmbH, Dessau
  - Nycomed Deutschland GmbH, Dierdorf
  - Nycomed Deutschland GmbH, Dillingen
  - Nycomed Deutschland GmbH, Dillingen-Diefflen
  - Nycomed Deutschland GmbH, Dinslaken
  - Nycomed Deutschland GmbH, Dorsten
  - Nycomed Deutschland GmbH, Dortmund
  - Nycomed Deutschland GmbH, Dörpen
  - Nycomed Deutschland GmbH, Dörzbach
  - Nycomed Deutschland GmbH, Dreetz
  - Nycomed Deutschland GmbH, Dresden
  - Nycomed Deutschland GmbH, Duisburg
  - Nycomed Deutschland GmbH, Dummerstorf
  - Nycomed Deutschland GmbH, Düren
  - Nycomed Deutschland GmbH, Dürrröhrsdorf
  - Nycomed Deutschland GmbH, Düsseldorf
  - Nycomed Deutschland GmbH, Ebeleben
  - Nycomed Deutschland GmbH, Ebersbach
  - Nycomed Deutschland GmbH, Eggenstein
  - Nycomed Deutschland GmbH, Ehingen
  - Nycomed Deutschland GmbH, Eimsheim
  - Nycomed Deutschland GmbH, Einbeck
  - Nycomed Deutschland GmbH, Eisenfeld
  - Nycomed Deutschland GmbH, Eisenhüttenstadt
  - Nycomed Deutschland GmbH, Eisfeld
  - Nycomed Deutschland GmbH, Eiterfeld
  - Nycomed Deutschland GmbH, Ellerstadt
  - Nycomed Deutschland GmbH, Elmshorn
  - Nycomed Deutschland GmbH, Elsenfeld
  - Nycomed Deutschland GmbH, Emleben
  - Nycomed Deutschland GmbH, Emmendingen
  - Nycomed Deutschland GmbH, Emsdetten
  - Nycomed Deutschland GmbH, Engelskirchen-Ründeroth
  - Nycomed Deutschland GmbH, Eningen unter Achalm
  - Nycomed Deutschland GmbH, Enkenbach-Alsenborn
  - Nycomed Deutschland GmbH, Erfurt
  - Nycomed Deutschland GmbH, Eschelbronn
  - Nycomed Deutschland GmbH, Eschwege
  - Nycomed Deutschland GmbH, Essen
  - Nycomed Deutschland GmbH, Fehmarn
  - Nycomed Deutschland GmbH, Fehrbellin
  - Nycomed Deutschland GmbH, Feldafing
  - Nycomed Deutschland GmbH, Felsberg-Gensungen
  - Nycomed Deutschland GmbH, Finsterwalde
  - Nycomed Deutschland GmbH, Flensburg
  - Nycomed Deutschland GmbH, Flonheim
  - Nycomed Deutschland GmbH, Flöha
  - Nycomed Deutschland GmbH, Framersheim
  - Nycomed Deutschland GmbH, Frankenberg/Eder
  - Nycomed Deutschland GmbH, Frankenthal
  - Nycomed Deutschland GmbH, Frankfurt
  - Nycomed Deutschland GmbH, Freiburg im Breisgau
  - Nycomed Deutschland GmbH, Freinsheim
  - Nycomed Deutschland GmbH, Freising
  - Nycomed Deutschland GmbH, Freyung
  - Nycomed Deutschland GmbH, Friedersdorf
  - Nycomed Deutschland GmbH, Friedrichshafen
  - Nycomed Deutschland GmbH, Friedrichsthal
  - Nycomed Deutschland GmbH, Friesenheim
  - Nycomed Deutschland GmbH, Frohburg
  - Nycomed Deutschland GmbH, Fürstenstein
  - Nycomed Deutschland GmbH, Fürstenwalde
  - Nycomed Deutschland GmbH, Fürth
  - Nycomed Deutschland GmbH, Gebesee
  - Nycomed Deutschland GmbH, Gefell
  - Nycomed Deutschland GmbH, Geisenheim
  - Nycomed Deutschland GmbH, Gelnhausen
  - Nycomed Deutschland GmbH, Gelsenkirchen
  - Nycomed Deutschland GmbH, Georgsmarienhütte
  - Nycomed Deutschland GmbH, Gera
  - Nycomed Deutschland GmbH, Geretsried
  - Nycomed Deutschland GmbH, Germering
  - Nycomed Deutschland GmbH, Gernrode
  - Nycomed Deutschland GmbH, Gladbeck
  - Nycomed Deutschland GmbH, Gleichen
  - Nycomed Deutschland GmbH, Goslar
  - Nycomed Deutschland GmbH, Goßwitz
  - Nycomed Deutschland GmbH, Görlitz
  - Nycomed Deutschland GmbH, Göttingen
  - Nycomed Deutschland GmbH, Göttingen-Elliehausen
  - Nycomed Deutschland GmbH, Gräfinau-Angstedt
  - Nycomed Deutschland GmbH, Greifswald
  - Nycomed Deutschland GmbH, Greiz
  - Nycomed Deutschland GmbH, Grevenbroich
  - Nycomed Deutschland GmbH, Grevesmühlen
  - Nycomed Deutschland GmbH, Grimma
  - Nycomed Deutschland GmbH, Groitzsch
  - Nycomed Deutschland GmbH, Großaitingen
  - Nycomed Deutschland GmbH, Großefehn
  - Nycomed Deutschland GmbH, Großenehrich
  - Nycomed Deutschland GmbH, Großkorbetha
  - Nycomed Deutschland GmbH, Gröden
  - Nycomed Deutschland GmbH, Grömitz
  - Nycomed Deutschland GmbH, Gundelsheim
  - Nycomed Deutschland GmbH, Güstrow
  - Nycomed Deutschland GmbH, Gütersloh
  - Nycomed Deutschland GmbH, Hagenow
  - Nycomed Deutschland GmbH, Halbe
  - Nycomed Deutschland GmbH, Halberstadt
  - Nycomed Deutschland GmbH, Halle
  - Nycomed Deutschland GmbH, Hamburg
  - Nycomed Deutschland GmbH, Hamelin
  - Nycomed Deutschland GmbH, Hamm
  - Nycomed Deutschland GmbH, Hammelburg
  - Nycomed Deutschland GmbH, Hanover
  - Nycomed Deutschland GmbH, Harsefeld
  - Nycomed Deutschland GmbH, Harsenwinkel
  - Nycomed Deutschland GmbH, Harsewinkel
  - Nycomed Deutschland GmbH, Hartenholm
  - Nycomed Deutschland GmbH, Hartenstein
  - Nycomed Deutschland GmbH, Haunsheim
  - Nycomed Deutschland GmbH, Haßmersheim
  - Nycomed Deutschland GmbH, Heek
  - Nycomed Deutschland GmbH, Heide
  - Nycomed Deutschland GmbH, Heidelberg
  - Nycomed Deutschland GmbH, Heilbronn
  - Nycomed Deutschland GmbH, Heiligemhafen
  - Nycomed Deutschland GmbH, Helmstadt
  - Nycomed Deutschland GmbH, Henningsdorf
  - Nycomed Deutschland GmbH, Herbsleben
  - Nycomed Deutschland GmbH, Hermsdorf
  - Nycomed Deutschland GmbH, Herne
  - Nycomed Deutschland GmbH, Herrnhut
  - Nycomed Deutschland GmbH, Herzberg
  - Nycomed Deutschland GmbH, Herzlake
  - Nycomed Deutschland GmbH, Herzogenaurach
  - Nycomed Deutschland GmbH, Hettstedt
  - Nycomed Deutschland GmbH, Hilpoltstein
  - Nycomed Deutschland GmbH, Hirschberg
  - Nycomed Deutschland GmbH, Hockenheim
  - Nycomed Deutschland GmbH, Homburg
  - Nycomed Deutschland GmbH, Homburg/ Saar
  - Nycomed Deutschland GmbH, Hoppegarten
  - Nycomed Deutschland GmbH, Horb
  - Nycomed Deutschland GmbH, Hoyerswerda
  - Nycomed Deutschland GmbH, Ilsenburg
  - Nycomed Deutschland GmbH, Ingelheim
  - Nycomed Deutschland GmbH, Ingolstadt
  - Nycomed Deutschland GmbH, Iserlohn
  - Nycomed Deutschland GmbH, Itzehoe
  - Nycomed Deutschland GmbH, Jarmen
  - Nycomed Deutschland GmbH, Jena
  - Nycomed Deutschland GmbH, Joachimsthal
  - Nycomed Deutschland GmbH, Jockgrim
  - Nycomed Deutschland GmbH, Jüterbog
  - Nycomed Deutschland GmbH, Kamen
  - Nycomed Deutschland GmbH, Kamenz
  - Nycomed Deutschland GmbH, Kamp-Lintfort
  - Nycomed Deutschland GmbH, Kandern-Wollbach
  - Nycomed Deutschland GmbH, Kappeln
  - Nycomed Deutschland GmbH, Karlsruhe
  - Nycomed Deutschland GmbH, Kaufbeuren
  - Nycomed Deutschland GmbH, Kemnitz
  - Nycomed Deutschland GmbH, Kerpen
  - Nycomed Deutschland GmbH, Ketzerbachtal/OT Raußlitz
  - Nycomed Deutschland GmbH, Kirchberg
  - Nycomed Deutschland GmbH, Kirchheimbolanden
  - Nycomed Deutschland GmbH, Koblenz
  - Nycomed Deutschland GmbH, Kolitzheim
  - Nycomed Deutschland GmbH, Korntal
  - Nycomed Deutschland GmbH, Kornwestheim
  - Nycomed Deutschland GmbH, Koßdorf
  - Nycomed Deutschland GmbH, Köhra
  - Nycomed Deutschland GmbH, Kressbronn
  - Nycomed Deutschland GmbH, Krumpa
  - Nycomed Deutschland GmbH, Künzelsau
  - Nycomed Deutschland GmbH, L.-E.-Musberg
  - Nycomed Deutschland GmbH, Laatzen
  - Nycomed Deutschland GmbH, Lampertheim
  - Nycomed Deutschland GmbH, Landau
  - Nycomed Deutschland GmbH, Landsberg
  - Nycomed Deutschland GmbH, Langenhagen
  - Nycomed Deutschland GmbH, Laubach
  - Nycomed Deutschland GmbH, Lauf
  - Nycomed Deutschland GmbH, Lauingen
  - Nycomed Deutschland GmbH, Lauterbach
  - Nycomed Deutschland GmbH, Lebach
  - Nycomed Deutschland GmbH, Lebus
  - Nycomed Deutschland GmbH, Lehesten
  - Nycomed Deutschland GmbH, Leimen
  - Nycomed Deutschland GmbH, Leinefelde-Worbis
  - Nycomed Deutschland GmbH, Leingarten
  - Nycomed Deutschland GmbH, Leipheim
  - Nycomed Deutschland GmbH, Leipzig
  - Nycomed Deutschland GmbH, Leisnig
  - Nycomed Deutschland GmbH, Lemförde
  - Nycomed Deutschland GmbH, Lengerich
  - Nycomed Deutschland GmbH, Leubnitz
  - Nycomed Deutschland GmbH, Leutenberg
  - Nycomed Deutschland GmbH, Leverkusen
  - Nycomed Deutschland GmbH, Lichtentanne
  - Nycomed Deutschland GmbH, Lieberose
  - Nycomed Deutschland GmbH, Linnich
  - Nycomed Deutschland GmbH, Lippstadt
  - Nycomed Deutschland GmbH, Loerrach
  - Nycomed Deutschland GmbH, Lotte-Wersen
  - Nycomed Deutschland GmbH, Loxstedt
  - Nycomed Deutschland GmbH, Löhne
  - Nycomed Deutschland GmbH, Löwenberg
  - Nycomed Deutschland GmbH, Lubnjow
  - Nycomed Deutschland GmbH, Ludwigsburg
  - Nycomed Deutschland GmbH, Ludwigshafen
  - Nycomed Deutschland GmbH, Lüdenscheid
  - Nycomed Deutschland GmbH, Lühmannsdorf
  - Nycomed Deutschland GmbH, Lünen
  - Nycomed Deutschland GmbH, Machern
  - Nycomed Deutschland GmbH, Magdeburg
  - Nycomed Deutschland GmbH, Mainaschaff
  - Nycomed Deutschland GmbH, Maintal
  - Nycomed Deutschland GmbH, Mainz
  - Nycomed Deutschland GmbH, Mannheim
  - Nycomed Deutschland GmbH, Marburg
  - Nycomed Deutschland GmbH, Markneukirchen
  - Nycomed Deutschland GmbH, Marl
  - Nycomed Deutschland GmbH, Märkisch Buchholz
  - Nycomed Deutschland GmbH, Meckenbeuren
  - Nycomed Deutschland GmbH, Meckenheim
  - Nycomed Deutschland GmbH, Meißen
  - Nycomed Deutschland GmbH, Mendig
  - Nycomed Deutschland GmbH, Menteroda
  - Nycomed Deutschland GmbH, Merseburg
  - Nycomed Deutschland GmbH, Merzen
  - Nycomed Deutschland GmbH, Merzig
  - Nycomed Deutschland GmbH, Messkirch
  - Nycomed Deutschland GmbH, Mettlach
  - Nycomed Deutschland GmbH, Metzingen
  - Nycomed Deutschland GmbH, Meuselwitz
  - Nycomed Deutschland GmbH, Miesbach
  - Nycomed Deutschland GmbH, Minden
  - Nycomed Deutschland GmbH, Mittelherwigsdorf
  - Nycomed Deutschland GmbH, Mochenwangen
  - Nycomed Deutschland GmbH, Mönchengladbach
  - Nycomed Deutschland GmbH, Mudau
  - Nycomed Deutschland GmbH, Mücheln
  - Nycomed Deutschland GmbH, Mühlhausen
  - Nycomed Deutschland GmbH, Mühlheim
  - Nycomed Deutschland GmbH, Mühltroff
  - Nycomed Deutschland GmbH, Mülheim
  - Nycomed Deutschland GmbH, Müncheberg
  - Nycomed Deutschland GmbH, München
  - Nycomed Deutschland GmbH, Münchweiler
  - Nycomed Deutschland GmbH, Nagold-Hochdorf
  - Nycomed Deutschland GmbH, Naumburg
  - Nycomed Deutschland GmbH, Neckargemünd
  - Nycomed Deutschland GmbH, Neckartailfingen
  - Nycomed Deutschland GmbH, Nettersheim
  - Nycomed Deutschland GmbH, Neubrandenburg
  - Nycomed Deutschland GmbH, Neudietendorf
  - Nycomed Deutschland GmbH, Neuenkirchen-Vörden
  - Nycomed Deutschland GmbH, Neukirchen-Vluyn
  - Nycomed Deutschland GmbH, Neumünster
  - Nycomed Deutschland GmbH, Neuseußlitz
  - Nycomed Deutschland GmbH, Neuss
  - Nycomed Deutschland GmbH, Neustadt
  - Nycomed Deutschland GmbH, Neustadt an der Orla
  - Nycomed Deutschland GmbH, Neuwied
  - Nycomed Deutschland GmbH, Niederlehme
  - Nycomed Deutschland GmbH, Norderstedt
  - Nycomed Deutschland GmbH, Nordstemmen
  - Nycomed Deutschland GmbH, Nuremberg
  - Nycomed Deutschland GmbH, Oberhausen
  - Nycomed Deutschland GmbH, Oberkirch
  - Nycomed Deutschland GmbH, Oberursel
  - Nycomed Deutschland GmbH, Offenburg
  - Nycomed Deutschland GmbH, Oftersheim
  - Nycomed Deutschland GmbH, Oranienburg
  - Nycomed Deutschland GmbH, Osnabrück
  - Nycomed Deutschland GmbH, Ostbevern
  - Nycomed Deutschland GmbH, Osterhausen
  - Nycomed Deutschland GmbH, Osterode
  - Nycomed Deutschland GmbH, Ostrhauderfehn
  - Nycomed Deutschland GmbH, Östringen
  - Nycomed Deutschland GmbH, Paderborn
  - Nycomed Deutschland GmbH, Panschwitz-Kuckau
  - Nycomed Deutschland GmbH, Passau
  - Nycomed Deutschland GmbH, Peckelsheim
  - Nycomed Deutschland GmbH, Peine
  - Nycomed Deutschland GmbH, Peine-Vöhrum
  - Nycomed Deutschland GmbH, Penig
  - Nycomed Deutschland GmbH, Pfaffenhofen
  - Nycomed Deutschland GmbH, Pforzheim
  - Nycomed Deutschland GmbH, Pfullingen
  - Nycomed Deutschland GmbH, Pfungstadt
  - Nycomed Deutschland GmbH, Pirmasens
  - Nycomed Deutschland GmbH, Pirna
  - Nycomed Deutschland GmbH, Plauen
  - Nycomed Deutschland GmbH, Plön
  - Nycomed Deutschland GmbH, Pohlheim
  - Nycomed Deutschland GmbH, Polch
  - Nycomed Deutschland GmbH, Porta Westfalica
  - Nycomed Deutschland GmbH, Potsdam
  - Nycomed Deutschland GmbH, Pößneck
  - Nycomed Deutschland GmbH, Prausitz
  - Nycomed Deutschland GmbH, Preetz
  - Nycomed Deutschland GmbH, Pritzwalk
  - Nycomed Deutschland GmbH, Pullach
  - Nycomed Deutschland GmbH, Radeberg
  - Nycomed Deutschland GmbH, Radis
  - Nycomed Deutschland GmbH, Radolfzell
  - Nycomed Deutschland GmbH, Rain A. Lech
  - Nycomed Deutschland GmbH, Rain Am Lech
  - Nycomed Deutschland GmbH, Ransbach-Baumbach
  - Nycomed Deutschland GmbH, Rastatt
  - Nycomed Deutschland GmbH, Ravensburg
  - Nycomed Deutschland GmbH, Remscheid
  - Nycomed Deutschland GmbH, Rendsburg
  - Nycomed Deutschland GmbH, Reutlingen
  - Nycomed Deutschland GmbH, Rietz Neuendorf
  - Nycomed Deutschland GmbH, Rinteln
  - Nycomed Deutschland GmbH, Rohrberg
  - Nycomed Deutschland GmbH, Rosenfeld
  - Nycomed Deutschland GmbH, Rostock
  - Nycomed Deutschland GmbH, Rotenburg (Wümme)
  - Nycomed Deutschland GmbH, Rottenburg
  - Nycomed Deutschland GmbH, Rödental
  - Nycomed Deutschland GmbH, Rödermark
  - Nycomed Deutschland GmbH, Röhrmoos
  - Nycomed Deutschland GmbH, Röthenbach
  - Nycomed Deutschland GmbH, Ruhmannsfelden
  - Nycomed Deutschland GmbH, Rüdersdorf
  - Nycomed Deutschland GmbH, Rülzheim
  - Nycomed Deutschland GmbH, Rüsselsheim am Main
  - Nycomed Deutschland GmbH, Saalburg-Ebersdorf
  - Nycomed Deutschland GmbH, Saalfeld
  - Nycomed Deutschland GmbH, Saarbrücken
  - Nycomed Deutschland GmbH, Sachsenheim
  - Nycomed Deutschland GmbH, Saint Blasien
  - Nycomed Deutschland GmbH, Saint Georgen
  - Nycomed Deutschland GmbH, Salching
  - Nycomed Deutschland GmbH, Sand
  - Nycomed Deutschland GmbH, Sandesneben
  - Nycomed Deutschland GmbH, Sanitz
  - Nycomed Deutschland GmbH, Schkeuditz
  - Nycomed Deutschland GmbH, Schlier
  - Nycomed Deutschland GmbH, Schneverdingen
  - Nycomed Deutschland GmbH, Schönberg
  - Nycomed Deutschland GmbH, Schönwalde
  - Nycomed Deutschland GmbH, Schwabach
  - Nycomed Deutschland GmbH, Schwalmstadt
  - Nycomed Deutschland GmbH, Schwarmstedt
  - Nycomed Deutschland GmbH, Schwarzenberg
  - Nycomed Deutschland GmbH, Schwarzheide
  - Nycomed Deutschland GmbH, Schwäbisch Hall
  - Nycomed Deutschland GmbH, Schwedt
  - Nycomed Deutschland GmbH, Schweinfurt
  - Nycomed Deutschland GmbH, Schwerin
  - Nycomed Deutschland GmbH, Seelow
  - Nycomed Deutschland GmbH, Siegen
  - Nycomed Deutschland GmbH, Silberhausen
  - Nycomed Deutschland GmbH, Sindelfingen
  - Nycomed Deutschland GmbH, Sittensen
  - Nycomed Deutschland GmbH, Sonderhausen
  - Nycomed Deutschland GmbH, Sondeshausen
  - Nycomed Deutschland GmbH, Sonneberg
  - Nycomed Deutschland GmbH, Speicher
  - Nycomed Deutschland GmbH, Spremberg
  - Nycomed Deutschland GmbH, Springe
  - Nycomed Deutschland GmbH, St.Ingbert
  - Nycomed Deutschland GmbH, Stadthagen
  - Nycomed Deutschland GmbH, Staßfurt
  - Nycomed Deutschland GmbH, Steinfeld
  - Nycomed Deutschland GmbH, Steinfurt
  - Nycomed Deutschland GmbH, Steißlingen
  - Nycomed Deutschland GmbH, Stendal
  - Nycomed Deutschland GmbH, Stiege
  - Nycomed Deutschland GmbH, Stockach
  - Nycomed Deutschland GmbH, Stralsund
  - Nycomed Deutschland GmbH, Straubing
  - Nycomed Deutschland GmbH, Strausberg
  - Nycomed Deutschland GmbH, Straßkirchen
  - Nycomed Deutschland GmbH, Stuhr
  - Nycomed Deutschland GmbH, Stuttgart
  - Nycomed Deutschland GmbH, Suhl
  - Nycomed Deutschland GmbH, Sulingen
  - Nycomed Deutschland GmbH, Sulz-Glatt
  - Nycomed Deutschland GmbH, Sulzbach
  - Nycomed Deutschland GmbH, Sulzheim
  - Nycomed Deutschland GmbH, Sundern
  - Nycomed Deutschland GmbH, Tarp
  - Nycomed Deutschland GmbH, Teltow
  - Nycomed Deutschland GmbH, Tessin
  - Nycomed Deutschland GmbH, Themar
  - Nycomed Deutschland GmbH, Thurnau
  - Nycomed Deutschland GmbH, Timmendorfer Strand
  - Nycomed Deutschland GmbH, Traunreut
  - Nycomed Deutschland GmbH, Triebes
  - Nycomed Deutschland GmbH, Trier
  - Nycomed Deutschland GmbH, Trossingen
  - Nycomed Deutschland GmbH, Tummendorfer Strand
  - Nycomed Deutschland GmbH, Tübingen
  - Nycomed Deutschland GmbH, Ueckermünde
  - Nycomed Deutschland GmbH, Uedem
  - Nycomed Deutschland GmbH, Uelzen
  - Nycomed Deutschland GmbH, Ulm
  - Nycomed Deutschland GmbH, Unterhaching
  - Nycomed Deutschland GmbH, Unterkirnach
  - Nycomed Deutschland GmbH, Überauchen
  - Nycomed Deutschland GmbH, Überlingen
  - Nycomed Deutschland GmbH, Vallendar
  - Nycomed Deutschland GmbH, Varel
  - Nycomed Deutschland GmbH, Veilsdorf
  - Nycomed Deutschland GmbH, Velbert
  - Nycomed Deutschland GmbH, Veringenstadt
  - Nycomed Deutschland GmbH, Viersen
  - Nycomed Deutschland GmbH, Visselhövede
  - Nycomed Deutschland GmbH, Voerde
  - Nycomed Deutschland GmbH, Wain
  - Nycomed Deutschland GmbH, Waldbröhl
  - Nycomed Deutschland GmbH, Waldkirch
  - Nycomed Deutschland GmbH, Wallerfangen
  - Nycomed Deutschland GmbH, Wandlitz
  - Nycomed Deutschland GmbH, Wassenberg
  - Nycomed Deutschland GmbH, Wattenheim
  - Nycomed Deutschland GmbH, Weibern
  - Nycomed Deutschland GmbH, Weida
  - Nycomed Deutschland GmbH, Weiden
  - Nycomed Deutschland GmbH, Weinböhla
  - Nycomed Deutschland GmbH, Weinheim-Oberflockenbach
  - Nycomed Deutschland GmbH, Weisenheim
  - Nycomed Deutschland GmbH, Weißenfels
  - Nycomed Deutschland GmbH, Weißwasser
  - Nycomed Deutschland GmbH, Welver
  - Nycomed Deutschland GmbH, Wennigsen
  - Nycomed Deutschland GmbH, Wesselburen
  - Nycomed Deutschland GmbH, Wesseling
  - Nycomed Deutschland GmbH, Westerrönfeld
  - Nycomed Deutschland GmbH, Wettringen
  - Nycomed Deutschland GmbH, Wetzlar
  - Nycomed Deutschland GmbH, Wiehl
  - Nycomed Deutschland GmbH, Wiesbaden
  - Nycomed Deutschland GmbH, Wilhelmshaven
  - Nycomed Deutschland GmbH, Willebadessen-Peckelsheim
  - Nycomed Deutschland GmbH, Willich
  - Nycomed Deutschland GmbH, Winkelhaid
  - Nycomed Deutschland GmbH, Winsen
  - Nycomed Deutschland GmbH, Wismar
  - Nycomed Deutschland GmbH, Wittenburg
  - Nycomed Deutschland GmbH, Wolfsburg
  - Nycomed Deutschland GmbH, Wörrstadt
  - Nycomed Deutschland GmbH, Wörth
  - Nycomed Deutschland GmbH, Wriedel
  - Nycomed Deutschland GmbH, Wuppertal
  - Nycomed Deutschland GmbH, Wustermark
  - Nycomed Deutschland GmbH, Zarrentin
  - Nycomed Deutschland GmbH, Zeitz
  - Nycomed Deutschland GmbH, Zernitz
  - Nycomed Deutschland GmbH, Zschopau
  - Nycomed Deutschland GmbH, Zweibrücken
  - Nycomed Deutschland GmbH, Zwickau
  - Nycomed Deutschland GmbH, Zwönitz

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: All patients were evaluated, missing values were not imputed.
Groups:
- Pantoprazole: All patients enrolled
Period: Overall Study
Arm/Group | Pantoprazole
Started | 4188
Completed | 4180
Not Completed | 8

BASELINE CHARACTERISTICS:
Arm/Group | Pantoprazole
Number analyzed (Participants) | 4188
Age Continuous [Mean (Standard Deviation); unit: years] — The measured value is related to the number of 4125 subjects (= valid cases). This number differs from the overall number of baseline participants due to missing data for 63 subjects.
  years | 55.3 (14.82)
Sex/Gender, Customized [Number; unit: percentage of participants]
  Female | 47.6
  Male | 52.0
  Missing data | 0.4
Nicotine use [Number; unit: percentage of participants]
  Smoker | 36.7
  Non-smoker | 62.8
  Missing data | 0.4
Alcohol use [Number; unit: percentage of participants]
  Daily | 21.9
  Not daily | 77.4
  Missing data | 0.6
Drug abuse [Number; unit: percentage of participants]
  Drug abuse | 3.6
  No drug abuse | 95.5
  Missing data | 0.9
Indication for prescription of pantoprazole [Number; unit: percentage of participants]
  Long-term therapy and/or relapse prophylaxis | 39.8
  Acute reflux oesophagitis | 57.2
  Missing data | 3.0

OUTCOME MEASURES:

1. Primary Outcome: Reflux-associated Gastrointestinal Symptoms: Assessment of the Severity of Heartburn
Description: Physician's assessment on a scale with 1=none, 2=mild, 3=moderate, 4=severe
Time Frame: 14 days
Population: Patients included and treated with valid data at first and last visit (without imputation of missing values), intention to treat
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Pantoprazole: All patients with valid values at first and last visit
Arm/Group | Pantoprazole
Number analyzed (Participants) | 4155
units on a scale
  Start of therapy | 3.10 (0.80)
  End of study | 1.36 (0.52)

2. Primary Outcome: Reflux-associated Gastrointestinal Symptoms: Assessment of the Severity of Eructation/Sour Eructation
Description: Physician's assessment on a scale with 1=none, 2=mild, 3=moderate, 4=severe
Time Frame: 14 days
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pantoprazole
Number analyzed (Participants) | 4155
units on a scale
  Start of therapy | 2.75 (0.89)
  End of study | 1.30 (0.50)

3. Primary Outcome: Reflux-associated Gastrointestinal Symptoms: Assessment of the Severity of Painful Swallowing
Description: Physician's assessment on a scale with 1=none, 2=mild, 3=moderate, 4=severe
Time Frame: 14 days
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pantoprazole
Number analyzed (Participants) | 4127
units on a scale
  Start of therapy | 1.87 (0.93)
  End of study | 1.06 (0.24)

4. Primary Outcome: Assessment of Pantoprazole at Final Visit: Efficacy Regarding Reflux Symptoms
Description: Physician's assessment on a scale with 1=excellent, 2=good, 3=satisfactory, 4=not satisfactory
Time Frame: 14 days
Population: Patients included and treated with at least one application of pantoprazole (without imputation of missing values), intention to treat
Measure: Number; unit: percentage of participants
Groups:
- Pantoprazole: Patients included and treated with at least one application of pantoprazole
Arm/Group | Pantoprazole
Number analyzed (Participants) | 4188
percentage of participants
  Excellent | 79.0
  Good | 19.2
  Satisfactory | 1.2
  Not satisfactory | 0.1
  Missing data | 0.5

5. Secondary Outcome: Functional Dyspepsia Symptoms: Assessment of the Severity of Upper Abdominal Pain
Description: Physician's assessment on a scale with 1=none, 2=mild, 3=moderate, 4=severe
Time Frame: 14 days
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pantoprazole
Number analyzed (Participants) | 4129
units on a scale
  Start of therapy | 2.21 (0.90)
  End of study | 1.17 (0.40)

6. Secondary Outcome: Functional Dyspepsia Symptoms: Assessment of the Severity of Sensation of Fullness
Description: Physician's assessment on a scale with 1=none, 2=mild, 3=moderate, 4=severe
Time Frame: 14 days
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pantoprazole
Number analyzed (Participants) | 4122
units on a scale
  Start of therapy | 2.35 (0.95)
  End of study | 1.26 (0.50)

7. Secondary Outcome: Functional Dyspepsia Symptoms: Assessment of the Severity of Nausea
Description: Physician's assessment on a scale with 1=none, 2=mild, 3=moderate, 4=severe
Time Frame: 14 days
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pantoprazole
Number analyzed (Participants) | 4055
units on a scale
  Start of therapy | 1.75 (0.82)
  End of study | 1.07 (0.27)

8. Secondary Outcome: Assessment of Pantoprazole at Final Visit: Efficacy Regarding Dyspeptic Symptoms
Description: Physician's assessment on a scale with 1=excellent, 2=good, 3=satisfactory, 4=not satisfactory
Time Frame: 14 days
Population: as for outcome 4
Measure: Number; unit: percentage of participants
Arm/Group | Pantoprazole
Number analyzed (Participants) | 4188
percentage of participants
  Excellent | 67.3
  Good | 26.0
  Satisfactory | 2.2
  Not satisfactory | 0.4
  Missing data | 4.2

9. Secondary Outcome: Irritable Bowel Syndrome: Assessment of the Severity of Lower Abdominal Pain
Description: Physician's assessment on a scale with 1=none, 2=mild, 3=moderate, 4=severe
Time Frame: 14 days
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pantoprazole
Number analyzed (Participants) | 4099
units on a scale
  Start of therapy | 1.39 (0.70)
  End of study | 1.06 (0.25)

10. Secondary Outcome: Irritable Bowel Syndrome: Assessment of the Severity of Diarrhoea
Description: Physician's assessment on a scale with 1=none, 2=mild, 3=moderate, 4=severe
Time Frame: 14 days
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pantoprazole
Number analyzed (Participants) | 4087
units on a scale
  Start of therapy | 1.26 (0.58)
  End of study | 1.05 (0.25)

11. Secondary Outcome: Irritable Bowel Syndrome: Assessment of the Severity of Constipation
Description: Physician's assessment on a scale with 1=none, 2=mild, 3=moderate, 4=severe
Time Frame: 14 days
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pantoprazole
Number analyzed (Participants) | 4090
units on a scale
  Start of therapy | 1.19 (0.53)
  End of study | 1.06 (0.27)

12. Secondary Outcome: Assessment of Pantoprazole at Final Visit: Efficacy Regarding Irritable Bowel Syndrome
Description: Physician's assessment on a scale with 1=excellent, 2=good, 3=satisfactory, 4=not satisfactory
Time Frame: 14 days
Population: as for outcome 4
Measure: Number; unit: percentage of participants
Arm/Group | Pantoprazole
Number analyzed (Participants) | 4188
percentage of participants
  Excellent | 53.9
  Good | 25.1
  Satisfactory | 5.9
  Not satisfactory | 0.7
  Missing data | 14.4

13. Secondary Outcome: Assessment of the Tolerability of Pantoprazole at Final Visit
Description: Physician's assessment on a scale with 1=excellent, 2=good, 3=satisfactory, 4=not satisfactory
Time Frame: 14 days
Population: as for outcome 4
Measure: Number; unit: percentage of participants
Arm/Group | Pantoprazole
Number analyzed (Participants) | 4188
percentage of participants
  Excellent | 84.5
  Good | 14.3
  Satisfactory | 0.5
  Not satisfactory | 0.02
  Missing data | 0.7

ADVERSE EVENTS:
Time Frame: From first until last visit
Arm/Group | Pantoprazole
Serious Adverse Events (participants affected / at risk) | 2/4188
Other Adverse Events (participants affected / at risk) | 3/4188
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pantoprazole (N=4188)
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 0.02% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pantoprazole (N=4188)
Diarrhoea (Gastrointestinal disorders) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No